CLINICAL TRIAL: NCT05135962
Title: Leaf Expander Versus Hyrax Expander. A Multicenter, Prospective, Randomized Trial
Brief Title: Maxillary Expansion: Leaf Expander Versus Hyrax Expander
Acronym: LEAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Genova (Other)
Collaborators: University of Milan (Other); Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, ALESSANDRO UGOLINI, Assistant Professor, University of Genova
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Leaf Expander mRCT
Record Dates: First submitted 2021-10-04; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Maxillary Deficiency
Keywords: maxillary expansion; slow expansion; rapid expansion; leaf expander
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- RME (rapid expansion) (Active Comparator): Intervention orthodontic - maxillary expansion:
  maxillary expansion with RME expander anchored on second deciduous molars. Activation: 1/turn day. RME was kept on teeth as a passive retainer and removed after one year from its application.
  Interventions: Device: orthodontic - rapid maxillary expansion
- Leaf expander 450g (slow expansion) (Experimental): Intervention orthodontic - maxillary expansion: maxillary expansion with Leaf Expander appliance anchored on second deciduous molars Activation: The leaves are preactivated in the laboratory to deliver 3mm of expansion. Reactivation is performed in the office by 10 quarter-turns of the screw per month until expansion has been completed. After active expansion, the Leaf Expander was kept on teeth as a passive retainer and removed after one year from its application.
  Interventions: Device: orthodontic - slow maxillary expansion with leaf expander
- Leaf self-expander 450g (slow expansion) (Experimental): Intervention orthodontic - maxillary expansion: maxillary expansion with Leaf self Expander appliance anchored on second deciduous molars.
  Activation: self activation (preactivated). After active expansion the Leaf self expander was kept on teeth as a passive retainer and removed after one year from its application
  Interventions: Device: orthodontic - slow maxillary expansion with self leaf expander
- Leaf expander 900g (slow expansion) (Experimental): Intervention orthodontic - maxillary expansion: maxillary expansion with Leaf Leaf Expander appliance anchored on second deciduous molars.
  Activation: The leaves are preactivated in the laboratory to deliver 3mm of expansion. Reactivation is performed in the office by 15 quarter-turns of the screw per month until expansion has been completed. After active expansion the Leaf Expander was kept on teeth as a passive retainer and removed after one year from its application.
  Interventions: Device: orthodontic - slow maxillary expansion with leaf expander
- Leaf self-expander 900g (slow expansion) (Experimental): Intervention orthodontic - maxillary expansion: maxillary expansion with Leaf self Expander appliance anchored on second deciduous molars.
  Activation: self activation (preactivated). After active expansion the Leaf self expander was kept on teeth as a passive retainer and removed after one year from its application
  Interventions: Device: orthodontic - slow maxillary expansion with self leaf expander

INTERVENTIONS:
Device: orthodontic - rapid maxillary expansion — Rapid expansion: when RME was in situ, patients started the screw activation of one-quarter turn a day until overcorrection was achieved and RME was kept on teeth as a passive retainer and removed after one year from its application.
  Other Names: orthodontic - rapid palatal expansion
  Arms: RME (rapid expansion)
Device: orthodontic - slow maxillary expansion with leaf expander — Leaf expander: The screw delivers a maximum expansion of 6 or 9 mm by activating (compressing) the spring, which generates a light (450g or 900g) and constant force. The leaves are preactivated in the laboratory to deliver 3mm of expansion. Reactivation is performed in the office by 10 quarter-turns (leaf 450g) or 15 quarter-turns (leaf 900g) of the screw per month until expansion has been completed. After active expansion the Leaf Expander is maintained passively in place for retention period. Leaf expander was kept on teeth as a passive retainer and removed after one year from its application.
  Other Names: orthodontic - slow palatal expansion with leaf expander
  Arms: Leaf expander 450g (slow expansion); Leaf expander 900g (slow expansion)
Device: orthodontic - slow maxillary expansion with self leaf expander — Leaf self expander: similar to Leaf expander with no need for reactivation or patient compliance.
  Other Names: orthodontic - slow palatal expansion with self leaf expander
  Arms: Leaf self-expander 450g (slow expansion); Leaf self-expander 900g (slow expansion)

SUMMARY:
The aim of the current study was to evaluate maxillary and mandibular arch widths' response to five different appliances and clinical protocols (Rapid maxillary expander RME, Leaf Expander 450g, Leaf Expander 900g, Self-expander 450g, Self-expander 900g) for the correction of the maxillary deficiency.

DETAILED DESCRIPTION:
Maxillary expansion with fixed appliance is a well-known and consolidated practice in clinical orthodontics but current findings of "evidence-based dentistry" have not yet identified a better clinical expansion protocol. This issue is due both to the several expansion screws available on the market and to the different screw activation protocols, which could be grouped in rapid and slow, with several customizations. The comparison between slow and rapid expansion is a hotly debated topic in the literature and a recent systematic review have shown that both rapid and slow expansion protocols are clinically effective on the primary outcome (the resolution of the maxillary deficiency and crossbite with a significant increase of skeletal transversal maxillary dimension). Based on these results, the choice of appliance based on its ability to solve the maxillary constriction may not be any more the main selection criteria. The choice of the orthodontist should also be based on the timing and on a "patient-oriented" device, that minimizes the side effects, such as e.g. appliance breakages, functional impairments, and pain perception.

The aim of the present study is to investigate and analyze five different maxillary expansion appliances to identify an effective and efficient clinical protocol for the maxillary expansion.

ELIGIBILITY:
Inclusion Criteria:

* prepubertal phase of development (cervical stage CS1 or 2 in cervical vertebral maturation or corresponding stage of third Finger middle phalanx maturation index).
* early or intermediate mixed dentition stage with fully erupted upper and lower first permanent molars.
* presence of the second upper deciduous molars available as an anchoring tooth. The second deciduous molar was considered available as anchoring tooth when the root had the same length as the clinical crown at the radiographic examination (Quinzi V, Federici Canova F, Rizzo FA, Marzo G, Rosa M, Primozic J. Factors related to maxillary expander loss due to anchoring deciduous molars exfoliation during treatment in the mixed dentition phase. Eur J Orthod. 2021 Jun 8;43(3):332-337. doi: 10.1093/ejo/cjaa061)
* Posterior transverse interarch discrepancy (PTID) of at least 3 mm. PTID was calculated on dental casts with a caliper as the difference between the maxillary intermolar width (distance between the central fossae of right and left permanent first maxillary molars) and the mandibular intermolar width (distance between the tips of the distobuccal cusps of right and left permanent first mandibular molars) (Tollaro, I., Baccetti, T., Franchi, L. and Tanasescu, C.D. 1996 Role of posterior transverse interarch discrepancy in Class II, Division 1 malocclusion during the mixed dentition phase. AJODO, 110, 417-422).

Exclusion Criteria:

* age older than 12 years,
* pubertal or postpubertal stage of development (CS 3-6),
* late deciduous or late mixed dentition, 4. agenesis of upper second premolars (assessed on initial panoramic radiograph),
* Class III malocclusion,
* cleft lip and/or palate and craniofacial syndromes

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Crossbite and/or traversal maxillary deficiency correction | 6 months
  Crossbite and/or traversal maxillary deficiency correction

SECONDARY OUTCOMES:
Crossbite correction stability | 1 year
  Crossbite correction stability
Crossbite correction stability | 2 years
  Crossbite correction stability
Canine and molar expansion (upper and lower arch) | 6 months
  Canine and molar millimetres of expansion (upper and lower arch)
Canine and molar angulation (upper and lower arch) | 6 months
  Canine and molar degrees of angulation (upper and lower arch)
Canine and molar expansion (upper and lower arch) | 1 year
  Canine and molar millimetres of expansion (upper and lower arch)
Canine and molar angulation (upper and lower arch) | 1 year
  Canine and molar degrees of angulation (upper and lower arch)
Upper and lower dental arch perimeter modifications | 6 months
  Upper and lower dental arch perimeter modifications (millimetres)
Upper and lower dental arch perimeter modifications | 1 year
  Upper and lower dental arch perimeter modifications (millimetres)
Pain during active expansion phase (VAS scale) | 1 month
  Pain during active expansion phase (VAS scale)
Appliance breakages and detachments | 6 months
  Appliance breakages and detachments
Number of in-office appointments | 6 months
  Number of in-office appointments
Time needed to correct the malocclusion | 6 months
  Time needed to correct the malocclusion

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Lanteri, DDS, Phd, Principal Investigator — University of Milan; Domenico Dalessandri, DDS, Phd, Principal Investigator — Università degli Studi di Brescia; Alessandro Ugolini, Principal Investigator — Universita degli Studi di Genova

REFERENCES:
- [Derived] Abate A, Ugolini A, Bruni A, Quinzi V, Lanteri V. Three-dimensional assessment on digital cast of spontaneous upper first molar distorotation after Ni-ti leaf springs expander and rapid maxillary expander: A two-centre randomized controlled trial. Orthod Craniofac Res. 2025 Feb;28(1):104-115. doi: 10.1111/ocr.12849. Epub 2024 Sep 8. PMID 39244736